CLINICAL TRIAL: NCT02837913
Title: Effect of a Warming Mattress on Perioperative Hypothermia Following Cesarean Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting study subjects
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Mark Zakowski MD, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00039382
Record Dates: First submitted 2016-07-06; First posted 2016-07-20 (Estimated); Results first posted 2018-10-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Hypothermia
Keywords: Perioperative Warming

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Underbody warmer on (Experimental): Underbody warmer will be underneath the patient and turned on.
  Interventions: Device: VitaHeat underbody heating mattress
- Underbody warmer off (Placebo Comparator): Underbody warmer will be underneath the patient but not turned on.
  Interventions: Device: VitaHeat underbody heating mattress

INTERVENTIONS:
Device: VitaHeat underbody heating mattress — Use of VitaHeat underbody heating mattress will be used for the intervention arm to reduce hypothermia post operatively

SUMMARY:
The primary aim of the current study will be to determine if the use of an underbody heating mattress during cesarean sections will decrease the incidence of postoperative hypothermia, defined as core temperature less than 36C, and if hypothermia occurs, time to normothermia. As part of the primary outcome the difference in the incidence of shivering, its severity, and need for treatment will be investigated. As a secondary goal other maternal perioperative outcomes will be studied i.e. estimated blood loss, change in hemoglobin level on the morning after surgery ie postop day 1, need for blood transfusion, rate of wound infections, length of hospital stay, maternal satisfaction, time to first breastfeeding, time to first 'skin to skin' contact. The relationship between maternal hypothermia and newborn outcomes of temperature and APGAR scores will also be evaluated.

Active preoperative and intraoperative warming may prevents inadvertent perioperative hypothermia and may be beneficial for pregnant patients undergoing cesarean delivery. The underbody warming mattress may be a step towards finding a suitable form of warming that is comfortable for awake patients, does not interfere with skin to skin contact and maternal-fetal bonding.

ELIGIBILITY:
Inclusion Criteria:

* will be age >18 years,
* singleton pregnancy >37 weeks,
* neuraxial anesthesia,
* healthy afebrile patients.

Exclusion Criteria:

* • will be age >18 years,

  * singleton pregnancy >37 weeks,
  * neuraxial anesthesia,
  * healthy afebrile patients.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Underbody Warmer on | Underbody Warmer Off
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Underbody Warmer on | Underbody Warmer Off | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (3.1) | 33.2 (5.6) | 34.6 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.1 (4.3) | 31.5 (7.4) | 29.2 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Temperature
Description: Temperature at time of post anesthesia care unit admission
Time Frame: 15 minute intervals until normothermic, up to 45 minutes after admission Post Anesthesia Care Unit
Measure: Mean (Standard Deviation); unit: Degrees Fahrenheit
Arm/Group | Underbody Warmer on | Underbody Warmer Off
Number analyzed (Participants) | 10 | 9
Degrees Fahrenheit
  Post Anesthesia Care Unit Admission | 96.5 (0.8) | 97.1 (0.8)
  15 minutes after admission | 96.0 (0.6) | 96.1 (1.0)
  30 minutes after admission | 96.7 (0.8) | 97.5 (0.7)
  45 minutes after admission | 96.9 (0.6) | 97.1 (0.8)

2. Secondary Outcome: Number of Participants With Shivering
Description: Shivering at time of post anesthesia care unit admission
Time Frame: 15 minute intervals until no shivering, up to 45 minutes after admission Post Anesthesia Care Unit
Measure: Count of Participants; unit: Participants
Arm/Group | Underbody Warmer on | Underbody Warmer Off
Number analyzed (Participants) | 10 | 9
Participants
  Arrival in post anesthesia care unit | 2 | 1
  15 minutes after admission | 2 | 0
  30 minutes after admission | 1 | 0
  45 minutes after admission | 0 | 0

3. Secondary Outcome: Vitals: Heart Rate
Description: Vitals: Heart Rate from preoperative through end of post anesthesia recovery unit
Time Frame: Preop up to 45 minutes after admission Post Anesthesia Care Unit, 15 min intervals
Population: healthy women undergoing cesarean
Measure: Mean (Standard Deviation); unit: beats per minutes
Arm/Group | Underbody Warmer on | Underbody Warmer Off
Number analyzed (Participants) | 10 | 9
beats per minutes
  Preoperative heart rate | 80.4 (10.3) | 77.1 (11.9)
  PostAnesthesia heart rate | 84.6 (12.8) | 79.8 (16.7)
  Delivery heart rate | 87.6 (13.8) | 80 (13.2)
  PostAnesthesiaRecoveryUnit Heart Rate Arrival | 89.4 (10.2) | 77.7 (10.9)
  PostAnesthesiaRecoveryUnit Heart Rate 15 minutes | 81.25 (17.2) | 62.5 (13.4)
  PostAnesthesiaRecoveryUnit Heart Rate 30 minutes | 81.5 (16.8) | 53 (0)
  PostAnesthesiaRecoveryUnit Heart Rate 45 minutes | 93 (0) | 53 (0)

4. Secondary Outcome: Blood Loss
Description: Estimated blood loss with and without warming
Time Frame: Documented at the end of 2 hour surgical procedure
Population: healthy pregnant women undergoing cesarean
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Underbody Warmer on | Underbody Warmer Off
Number analyzed (Participants) | 10 | 9
milliliter | 630 (143.76) | 711.11 (170.99)

5. Secondary Outcome: Time to Neonatal Bonding
Description: time to neonatal bonding as skin to skin
Time Frame: time from delivery to first maternal contact during the 2 hour surgical procedure
Population: healthy women undergoing cesarean
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Underbody Warmer on | Underbody Warmer Off
Number analyzed (Participants) | 10 | 9
minutes | 32 (29) | 13 (10.3)

6. Secondary Outcome: Thermal Comfort Visual Analog Scale
Description: Thermal comfort visual analog scale with scores 0-100 with 50 being temperature comfort/neutral, 100 being hottest, 0 being cold
Time Frame: Preop up to 45 minutes after admission Post Anesthesia Care Unit, 15 min intervals
Population: health women undergoing cesarean
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Underbody Warmer on | Underbody Warmer Off
Number analyzed (Participants) | 10 | 9
units on a scale
  Preoperative thermal comfort | 50.8 (3.3) | 48.9 (4.2)
  PostAnesthesia thermal comfort | 48.5 (3.4) | 47.8 (3.6)
  Delivery Thermal Comfort | 49.5 (1.6) | 46.1 (4.9)
  PostAnesthesiaRecoveryUnit Thermal Comfort Arrival | 49.5 (3.7) | 45.6 (9.2)
  PostAnesthesiaRecoveryUnit Thermal Comfort 15 min | 46.3 (4.8) | 50 (0)
  PostAnesthesiaRecoveryUnit Thermal Comfort 30 min | 47.5 (5) | 50 (0)
  PostAnesthesiaRecoveryUnit Thermal Comfort 45 min | 50 (0) | 50 (0)

7. Secondary Outcome: Vitals: Oxygen Saturation
Description: Vitals: Oxygen Saturation from preoperative through end post anesthesia recovery unit
Time Frame: Preop up to 45 minutes after admission Post Anesthesia Care Unit, 15 min intervals
Population: healthy women undergoing cesarean
Measure: Mean (Standard Deviation); unit: oxygen saturation, %
Arm/Group | Underbody Warmer on | Underbody Warmer Off
Number analyzed (Participants) | 10 | 9
oxygen saturation, %
  Preoperative oxygen saturation | 99.8 (0.4) | 99.7 (1)
  postAnesthesia oxygen saturation | 98.8 (2.8) | 99.9 (0.3)
  Delivery oxygen saturation | 98.3 (1.3) | 99.1 (1.1)
  PostAnesthesiaRecoveryUnit OxygenSaturationArrival | 98.4 (1.6) | 98.7 (1.4)
  PostAnesthesiaRecoveryUnit OxygenSaturation15minut | 99.8 (0.5) | 99.5 (0.7)
  PostAnesthesiaRecoveryUnit OxygenSaturation30minut | 98.8 (1.3) | 99 (0)
  PostAnesthesiaRecoveryUnit OxygenSaturation45minut | 99 (0) | 99 (0)

8. Secondary Outcome: Vitals: Blood Pressure
Description: Vitals: blood pressure as mean arterial pressure
Time Frame: Preop up to 45 minutes after admission Post Anesthesia Care Unit, 15 min intervals
Population: healthy women undergoing cesarean
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Underbody Warmer on | Underbody Warmer Off
Number analyzed (Participants) | 10 | 9
mmHg
  Preoperative Blood Pressure | 92.9 (11) | 84.2 (6.7)
  PostAnesthesia Blood Pressure | 93.3 (12.9) | 90.5 (14.4)
  Delivery Blood Pressure | 84.4 (10.2) | 92.3 (8.9)
  PostAnesthesiaRecoveryUnit BloodPressure Arrival | 82.3 (15.3) | 77.1 (9.2)
  PostAnesthesiaRecoveryUnit BloodPressure 15minutes | 84.3 (12.1) | 85 (2.8)
  PostAnesthesiaRecoveryUnit BloodPressure 30minutes: number analyzed (Participants) | 10 | 0
  PostAnesthesiaRecoveryUnit BloodPressure 30minutes | 85.8 (12.8) |
  PostAnesthesiaRecoveryUnit BloodPressure 45minutes: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Underbody Warmer on | Underbody Warmer Off
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT02837913/Prot_SAP_001.pdf